CLINICAL TRIAL: NCT05315232
Title: Glanzmanns 360. The Lived Experience of People With Glanzmanns.
Brief Title: The Experiences of People Who Live With Glanzmanns Thrombasthenia.
Status: Completed | Type: Observational
Sponsor: Haemnet (Other)
Collaborators: Hemab ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: Glanzmanns 360
Record Dates: First submitted 2022-03-15; First posted 2022-04-07 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Glanzmann Thrombasthenia
MeSH Terms: conditions — Thrombasthenia | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Qualitative assessment: Survey (using validated quality of life assessment questionnaires) and one to one interviews of people and family members living with Glanzmanns Thrombasthenia
  Interventions: Other: survey and interview
- Bleed diary: Daily bleed diary completion over 12 weeks
  Interventions: Other: survey and interview

INTERVENTIONS:
Other: survey and interview — qualitative assessment
  Other Names: diary completion

SUMMARY:
To understand the lived experiences of people with Glanzmanns Thrombasthenia

DETAILED DESCRIPTION:
A qualitative study of people with Glanzmanns Thrombasthenia including an on-line survey, qualitative in-depth interviews and bleed diary completion.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of congenital (inherited) Glanzmanns Thrombasthenia

Exclusion Criteria:

Acquired Glanzmanns Thrombasthenia

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with Glanzmanns Thrombasthenia or parents of children with Glanzmanns Thrombasthenia.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
to understand the impact of GT on quality of life of affected individuals and their families. | one year
  Incidence of reported impact of GT on daily life using validated questionnaires EQ5D, MIQ, PHQ9, Rosenbergs self esteem scale.

SECONDARY OUTCOMES:
Identify levels of acceptability of current treatments and management approaches | one year
  Rate of reported satisfaction with current treatments using self efficacy to manage disease assessment tool
Identify areas of unmet need among people with GT | one year
  Rate of reported unmet need using ED5D and MIQ

CONTACTS AND LOCATIONS:
Overall Officials: Mike Holland, BSC, Study Director — Haemnet
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The second part of the study will be conducted by Haemnet and Hemab - participant information will be shared after reconsenting
Supporting Information: ICF, CSR
Time Frame: 3-6 months